CLINICAL TRIAL: NCT03222999
Title: Korean Cardiac Arrest Research Consortium
Status: Recruiting | Type: Observational
Sponsor: Korean Cardiac Arrest Research Consortium (Other)
Responsible Party: Principal Investigator, Chung, Sung-Phil, Study Chair, Korean Cardiac Arrest Research Consortium
Other Study IDs: KoCARC
Record Dates: First submitted 2017-07-06; First posted 2017-07-19 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: Out-of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention planned — No intervention planned

SUMMARY:
This study will evaluated the epidemiology and the outcomes of patients suffering out-of-hospital cardiac arrest with presumed cardiac etiology in Korea.

DETAILED DESCRIPTION:
The Korean Cardiac Arrest Research Consortium (KoCARC) is a collaborative research network developed to comprehend various researches conducted in the field of out-of-cardiac arrest resuscitation and to strengthen the cooperative effort in conducting studies. It was organized in 2014 with recruitment of hospitals willing to participate voluntarily to the consortium.

Not only for emergency medicine, but KoCARC is expanding the research collaboration with cardiology, preventive medicine and epidemiology as well. To enhance the professionalism and effectiveness in research, seven research committees, which consists of Epidemiology and Preventive Research Committee (EPR), Community Resuscitation Research Committee (CRR), EMS Resuscitation Research Committee (ERR), Hospital Resuscitation Research Committee (HRR), Hypothermia and Post-resuscitation Care Research Committee (HPR), Cardiac Care Resuscitation Committee (CCR) and Pediatric Resuscitation Research Committee (PRR). Also Data Safety and Monitoring Board Committee (DSMB) is organized to provide annual review and Security and Ethics Committee to oversight security and ethical issues in research. Monthly meeting of interdisciplinary steering committee, consists of the consortium chair, steering committee chair, each research committee chair and secretary committee, is held to approve the proposed research agendas and to mediate between multi-center trial participating hospitals.

KoCARC registry is a data collecting system composed of OHCA risk and prognostic variables developed to provide the platform to researches conducted in KoCARC.

ELIGIBILITY:
Inclusion Criteria:

* OHCA patients who were transported to participating emergency department (ED) by emergency medical service with resuscitation efforts and whose arrest was identified as a presumed cardiac etiology by emergency physicians in ED.

Exclusion Criteria:

* OHCA with terminal illness documented by medical record, under hospice care, with pregnancy, with pre-documented 'Do Not Resuscitate' card
* OHCA of definite non-cardiac etiology, including trauma, drowning, poisoning, burn, asphyxia, or hanging

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: EMS treated OHCA who visits study participating ED
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival at 6 month | 6 months after cardiac arrest
  Patients will be followed upon hospital discharge and up to 6 month.

SECONDARY OUTCOMES:
Good neurological recovery at 6 month | 6 months after cardiac arrest
  Good neurological recovery: Cerebral Performance Category (CPC) 1 or 2. Patients will be followed upon hospital discharge and up to 6 month.

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Pil Chung, MD, PhD, Study Chair — Korean Cardiac Arrest Resuscitation Consortium
Locations (1):
- Korean Cardiac Arrest Resuscitation Consortium, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi A, Park I, You JS, Chung SP, Park YS. Non-Linear Relationship Between Alcohol Consumption and Neurological Outcomes in Patients With Out-of-Hospital Cardiac Arrest Presenting to the Emergency Department. J Korean Med Sci. 2025 Jun 2;40(21):e96. doi: 10.3346/jkms.2025.40.e96. PMID 40461141
- [Derived] Lee H, Oh J, Choi HJ, Shin H, Cho Y, Lee J. The Incidence and Outcomes of Out-of-Hospital Cardiac Arrest During the COVID-19 Pandemic in South Korea: Multicenter Registry Study. JMIR Public Health Surveill. 2024 Jun 24;10:e52402. doi: 10.2196/52402. PMID 38913998
- [Derived] Ko BS, Kim YJ, Han KS, Jo YH, Shin J, Park I, Kang H, Lim TH, Hwang SO, Kim WY. Association between the number of prehospital defibrillation attempts and a sustained return of spontaneous circulation: a retrospective, multicentre, registry-based study. Emerg Med J. 2023 Jun;40(6):424-430. doi: 10.1136/emermed-2021-212091. Epub 2023 Apr 6. PMID 37024298
- [Derived] Jeong D, Lee GT, Park JE, Chang H, Kim T, Cha WC, Yoon H, Hwang SY, Shin TG, Sim MS, Jo I, Lee SH, Shin SD, Choi JH. Extracorporeal Life-support for Out-of-hospital Cardiac Arrest: A Nationwide Multicenter Study. Shock. 2022 May 1;57(5):680-686. doi: 10.1097/SHK.0000000000001924. Epub 2022 Mar 10. PMID 35271541
- [Derived] Kim SJ, Kim HS, Hwang SO, Jung WJ, Roh YI, Cha KC, Shin SD, Song KJ; Korean Cardiac Arrest Research Consortium (KoCARC) Investigators. Ionized calcium level at emergency department arrival is associated with return of spontaneous circulation in out-of-hospital cardiac arrest. PLoS One. 2020 Oct 12;15(10):e0240420. doi: 10.1371/journal.pone.0240420. eCollection 2020. PMID 33045006
- [Derived] Yoon JC, Kim YJ, Ahn S, Jin YH, Lee SW, Song KJ, Shin SD, Hwang SO, Kim WY; Korean Cardiac Arrest Research Consortium KoCARC. Factors for modifying the termination of resuscitation rule in out-of-hospital cardiac arrest. Am Heart J. 2019 Jul;213:73-80. doi: 10.1016/j.ahj.2019.04.003. Epub 2019 May 3. PMID 31129440
- [Derived] Lee DE, Lee MJ, Ahn JY, Ryoo HW, Park J, Kim WY, Shin SD, Hwang SO; Korean Cardiac Arrest Research Consortium (KoCARC). New Termination-of-Resuscitation Models and Prognostication in Out-of-Hospital Cardiac Arrest Using Electrocardiogram Rhythms Documented in the Field and the Emergency Department. J Korean Med Sci. 2019 May 6;34(17):e134. doi: 10.3346/jkms.2019.34.e134. PMID 31050224